CLINICAL TRIAL: NCT04476888
Title: Convalescent Plasma Treatment in COVID-19 Patients at a Tertiary Care Center in Pakistan
Brief Title: Convalescent Plasma Treatment in COVID-19
Acronym: COLLATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Muhammad Hasan, Senior Instructor, Aga Khan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CON000000000880
Record Dates: First submitted 2020-07-16; First posted 2020-07-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Covid19
Keywords: Convalescent plasma; Covid 19
MeSH Terms: conditions — COVID-19 | interventions — Pharmaceutical Preparations; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm/CP recipient (Experimental): Patients with severe/critical COVID 19 who will receive 500 ml of Convalescent plasma (CP), obtained from donors who have been recovered from SARS-CoV-2 infection.
  These patients may or may not get other treatment modalities e.g. steroids,Tocilizumab, Azithromycin etc
  Interventions: Biological: Convalescent Plasma (CP); Other: Drugs and supportive care
- Control arm (Other): Patients with severe/critical COVID 19 who will not receive Convalescent plasma (CP). These will be those who were recruited during the period before CP becomes available or for whom no compatible CP is available.
  These patients will receive one or more of the other treatment modalities e.g. steroids,Tocilizumab, Azithromycin etc
  Interventions: Other: Drugs and supportive care

INTERVENTIONS:
Biological: Convalescent Plasma (CP) — 500 ml of Convalescent plasma in a single dose will be transfused over a period of 1- 2 hours.
  Arms: Treatment arm/CP recipient
Other: Drugs and supportive care — This will include drugs like steroids, tocilizumab, azithromycin and supportive care

SUMMARY:
The outbreak of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) occurred initially in December 2019 in the city of Wuhan, Hubei province, China. Patients mainly presented with respiratory symptoms and this novel pathogen was identified.At present, the core management of COVID-19 includes infection prevention, case detection, monitoring, and supportive care. While specific new drugs and vaccines are being researched, certain drugs that are already present in medical arsenal are under trial too.

One investigational treatment being explored for COVID-19 is the use of convalescent plasma (CP) collected from recovered COVID-19 patients. Convalescent Plasma is a source of passive immune therapy- the administration of specific antibodies against a given agent for preventing or treating an infectious disease due to that agent. The main anticipated mechanism of action of Convalescent Plasma therapy in COVID19 is viral neutralization. Other possible mechanisms include antibody-dependent cellular cytotoxicity and phagocytosis. There are numerous examples in which convalescent plasma (CP) has been used successfully as post exposure prophylaxis and/or treatment of infectious diseases, including other outbreaks of coronaviruses e.g. SARS-1, MERS-CoV and very recently in 2014, the Ebola virus outbreak. In SARS-CoV-2, Shen et al published a case series of 5 critically ill patients with COVID-19 and acute respiratory distress syndrome showing improvement in clinical status after transfusion of CP.

Therefore, the objective of this study is to determine the safety and efficacy of transfusing convalescent plasma in patients admitted with COVID-19 at Aga Khan University Karachi, Pakistan. The investigators hypothesize that CP will decrease the length of hospital stay and overall mortality in patients with COVID-19.

In this study, convalescent plasma will be collected from the donors who have been recovered from SARS-CoV-2 infection and transfused it to the patients admitted with active severe /critical COVID-19 at the Aga Khan University Hospital Karachi.

STUDY DESIGN: Non-randomized open Label trial

INCLUSION CRITERIA IN TREATMENT ARM:

i. Inpatients at AKU with positive SARS-CoV-2 infection by rRT-PCR and who have provided written informed consent for inclusion in the trial;

ii. Age ≥ 18 years;

iii. Severe or immediately life-threatening COVID-19 defined by any of:

* Respiratory rate ≥ 30/min;
* Blood oxygen saturation ≤ 93% at room air;
* Partial pressure of arterial Oxygen to Fraction of inspired Oxygen ratio < 300;
* Lung infiltrates > 50% within 24 to 48 hours on radiology ( X-ray or CT scan);
* Need for mechanical ventilation.
* respiratory failure
* septic shock
* multiple organ dysfunction or failure

EXCLUSION CRITERIA:

i. Negative rRT-PCR from respiratory secretions or blood within 48 h prior to assessment of eligibility.

ii. History of allergic reaction to blood or plasma products (as judged by the investigator).

iii. Medical conditions in which receipt of 500 mL intravascular volume may be detrimental to the patient (e.g., actively decompensated congestive heart failure).

iv. Enrolment in any other clinical trial for an investigational therapy.

CONTROL GROUP:

COVID-19 patients recruited during the period before CP becomes available or for whom no compatible CP is available will be given Standard of Care and will be followed for study outcomes. Data from these SC patients will be used as comparator in the analysis of the study.

DETAILED DESCRIPTION:
Objective:

To investigate the efficacy and safety of transfusing convalescent plasma collected from patients who have recovered from COVID-19 disease to patients admitted at Aga Khan University Hospital for the management of active COVID-19 disease.

Methods:

A. Study design Non-randomized open Label trial

B. Study population

1. CP donors:

   Inclusion criteria: All the following should be met:

   i. Outpatients or discharged inpatients of AKUH diagnosed with SARS-CoV-2 infection by real time Reverse Transcriptase-Polymerase Chain Reaction (rRT-PCR) and who have provided written informed consent for inclusion in the trial; ii. Evidence of viral clearance by negative rRT-PCR at (1) clinical recovery and (2) 24 hours before the intended time of CP collection. The interval between these two tests should be at least 14 days.

   iii. Age between 18- 60 years

   Exclusion criteria Ineligible to donate plasma according to donor selection criteria used at AKUH blood bank

   CP recipients (treatment arm):

   Inclusion criteria i. Inpatients at AKU with positive SARS-CoV-2 infection by rRT-PCR and who have provided written informed consent for inclusion in the trial; ii. Age ≥ 18 years; iii. Severe or immediately life-threatening COVID-19 defined by any of:
   * Respiratory rate ≥ 30/min;
   * Blood oxygen saturation ≤ 93% at room air;
   * Partial pressure of arterial Oxygen to Fraction of inspired Oxygen ratio < 300;
   * Lung infiltrates > 50% within 24 to 48 hours on radiology ( X-ray or CT scan);
   * Need for mechanical ventilation.
   * respiratory failure
   * septic shock
   * multiple organ dysfunction or failure

   Exclusion criteria i. Negative rRT-PCR from respiratory secretions or blood within 48 h prior to assessment of eligibility.

   ii. History of allergic reaction to blood or plasma products (as judged by the investigator).

   iii. Medical conditions in which receipt of 500 mL intravascular volume may be detrimental to the patient (e.g., actively decompensated congestive heart failure).

   iv. Enrolment in any other clinical trial for an investigational therapy.
2. Control group:

COVID-19 patients recruited during the period before CP becomes available or for whom no compatible CP is available will be given Standard of Care and will be followed for study outcomes. Data from these SC patients will be the used as comparator in the analysis of the study.

C. Informed consent

1. CP donors: Consent for CP donation from those eligible to donate will be taken by the principal investigator.
2. CP recipient: Informed consent will be taken by a healthcare provider in the primary team caring for the patient using standard infection control precautions. If the patient is deemed to lack capacity for consent, then consent will be taken by next of kin.

D. Study procedures

1. Convalescent Plasma Collection and Storage:

   Potential donors who meet the inclusion criteria and have given informed consent will undergo pre-donation testing to assess final suitability for donation, according to the routine policy and procedures. Pre-donation testing will include:
   * ABO and RhD grouping
   * Blood screening tests for transfusion transmissible infections according to the blood bank routine policy and procedures including serology of HBV, HCV, HIV, malaria & syphilis and nucleic acid testing (NAT) for HBV, HCV and HIV.
   * IgG antibody testing through SARS-CoV-2 IgG antibodies ELISA Kits (Sample will also be stored for PRNT testing which will be performed later when facility become available) The results of pre-donation testing will be reviewed. Potential donors who test negative for all TTI tests and positive for SARS CoV-2 Ig G antibodies, will be selected for CP donations. CP will preferably be collected by apheresis from donors as it enables collection and storage of large volumes of CP that may be used for more than one patient. In apheresis procedure, approximately one-liter plasma would be obtained from the donor and replacement fluid (1000ml normal saline) will be infused. This 1000 ml plasma will be divided into 2 portions of 500 ml each, so that it can be used to transfuse 2 patients.

   Principle of Apheresis : Donor apheresis is a process in which whole blood is withdrawn from a donor's circulation; desired component (platelets, plasma, red blood cells or stem cells) is separated out and retained while remainder is returned to the donor. During apheresis the blood pumps through the cell-separator and the desired components are collected in a sterile plastic container and recombined remaining elements are returned to the donor.

   Pre-procedural steps:
   * Ensure donor identity.
   * Ensure that the donor has had something to eat and drink prior to apheresis.
   * Measure and record weight and height.
   * On-call doctor ensures the donor is fit to undergo the procedure.
   * Doctor fills donor assessment form before procedure and technologist also fill remaining column of assessment form during and after procedure.
   * Inform consent is obtained by medical doctor and signed by donor with all risks discussed.

   Procedure:

   The apheresis technologist installs kit and primes the machine for the procedure as per manufacturer's guidelines or manual. Then he enters the donor's age, gender, weight, height, and hematocrit in a machine. Then machine displays total blood volume.

   When machine is ready, technologist cleans the insides of both arms; inserts a needle into one vein in each arm, connects the donor to the apheresis machine. Performs procedure as per manufactures manual. Blood is drawn from one of the donor's arms and is spun in a centrifuge within the machine thus separating platelets from whole blood. The donor's blood is in a sterile, closed-system apheresis kit within centrifuge. This kit allows the blood to be spun in the centrifuge and prevent it from touching the machine, eliminating the risk of contamination. After the plasma separation, the donor's red cells, white cells and platelets return to the donor through the other arm.

   When the desired component collected select reinfusion and the blood remaining in the circuit is returned to the donor. Needles are the removed and pressure is applied to the venipuncture site until bleeding has stopped. A pressure dressing is then applied to the phlebotomy site. Kit and other disposable items dispose-off in an appropriate biohazard disposable container and send for incineration.

   When procedure is completed, post-donation instructions are given to donor, and after procedure technologist asks the donor to rest for15 to 20 minutes (written information at time of donation).

   If donor is feeling well, he/she asked to stand by the chair for a few moments to ensure that do not experience hypotension. Otherwise see a doctor if feels uncomfortable.

   The donor would be provided with good care before, during and after the whole blood donation or apheresis procedure. On-call doctor and medical technologist will monitors donor throughout procedure. Any adverse donor reactions will be adequately and promptly managed and recorded as per routine blood bank policy and procedures.

   The inter-donation interval for collection of plasma by apheresis would be no less than two weeks.

   Only if a donor is not fit to undergo apheresis or does not agree for the apheresis procedure, then such donor will be given the option to donate Whole Blood. This method will be just like routine blood donation in which we will collect 450-500 ml whole blood from the donor in a bag. We will then use the collected whole blood bag to prepare plasma (approx. 150 ml plasma) by centrifugation, as per routine blood bank SOP. The plasma collected by this whole blood method will need pooling i.e. 3 plasma units collected from different donors will be pooled to get a single patient's dose (500 ml).

   Potential donors with abnormal TTI test results would not be accepted and will be referred to appropriate health-care institutions for further investigation, confirmation, counselling, treatment and care.

   CP separated from whole blood donations or collected by apheresis will be stored as 'liquid plasma' between +2 degree centigrade and +6 degree centigrade in blood bank refrigerators for up to 40 days. Alternatively, it will be frozen either within 8 hours of collection as 'Fresh Frozen Plasma' or within 18-24 hours of collection as 'Plasma Frozen Within 24 hours' and stored for up to 12 months at or below -18 degree centigrade in a controlled plasma freezer.
2. Administration of Convalescent Plasma therapy to patients COVID-19 patients who meet the eligibility criteria for treatment will be approached for consent.

Patients will have their blood type determined. CP must be ABO compatible with the recipient's blood type.

Whether plasma have been obtained from apheresis procedure or separated from whole blood donation, the transfusion protocol would be the same. Patients will receive two consecutive transfusions of 250 ml of ABO-compatible convalescent plasma (i.e. 500 ml of convalescent plasma in total). Each transfusion will be administered over a 20-minute period, with a 15-minute interval between the two transfusions. Transfusion will be done in accordance with the standard policy routinely used at hospital for administration of blood products.

E. Concomitant therapy The clinical team will have complete independent control of patient management and as such, management other than CP therapy will not be influenced by the intervention or study team. Co-interventions, including corticosteroids, antiviral drugs, interferon etc. will be documented on the study case report forms.

F. Withdrawal of subjects Subjects may voluntarily withdraw from the trial at any time after informing the investigators. At the time of informed consent and again at communication of this decision, the importance of staying in the study for the full duration of follow-up will be explained to subjects by the investigators. The reason for withdrawal will be documented.

For subjects who withdraw due to adverse events (AEs) defined below, investigators will closely follow up their AEs until the subject returns to the baseline state or till their condition is stable. If subjects are lost to follow-up, existing data collected until the time of loss to follow up will be used for analysis.

Adverse events:

Slow intravenous transfusion of convalescent plasma therapy will be given with careful monitoring of the patient for any acute transfusion reactions, particularly during the first 15-20 minutes. Transfusion will be completed within 2 hours of commencement with monitoring and recording of the patient's vital signs by the transfusion nurse. Adverse events are defined as any serious or intolerable events which, in the investigators' judgement, requires withdrawal of the subject from the study. These include:

1. Allergic reactions (including oropharyngeal edema, severe rash, bronchospasm, and immediate-type allergic reactions).
2. Complications of intravascular volume overload and transfusion-related acute lung injury (TRALI).
3. Serious adverse events

   1. Life-threatening
   2. Death
   3. Significant disability/incapacity
   4. Hospitalization or prolonged hospitalization
   5. Congenital abnormality

Ethics The trial will be conducted in compliance with the principles of the Declaration of Helsinki (version 2013), and to principles of Good Clinical Practice. Inclusion in the trial will be voluntary and subject to provision of written informed consent. Each participant will be informed of their right to withdraw from the study at any time without penalty or loss of benefits including standard of care. Confidentiality of all subjects will be maintained throughout the trial. Blood and plasma units will be stored using ID numbers instead of identifiable information. Access to subject medical records will be provided to authorized staff only.

Ethical approval has been obtained from the AKUH ethics Review Committee and National Bioethics Committe before trial commencement and any subsequent protocol amendments will be submitted to the ERC immediately. A copy of the Final study report will also be submitted to the ERC.

PI will monitor data frequently for quality and completeness. CRF data will be derived from source data and all CRFs will be kept in lock and key. Electronic data will be stored in principal investigator's computer in a password protected file.

ELIGIBILITY:
Inclusion Criteria For Patients:

i. Inpatients at AKU with positive SARS-CoV-2 infection by rRT-PCR and who have provided written informed consent for inclusion in the trial;

ii. Age ≥ 18 years;

iii. Severe or immediately life-threatening COVID-19 defined by any of:

* Respiratory rate ≥ 30/min;
* Blood oxygen saturation ≤ 93% at room air;
* Partial pressure of arterial Oxygen to Fraction of inspired Oxygen ratio < 300;
* Lung infiltrates > 50% within 24 to 48 hours on radiology ( X-ray or CT scan);
* Need for mechanical ventilation.
* respiratory failure
* septic shock
* multiple organ dysfunction or failure

Exclusion Criteria for patients:

i. Negative rRT-PCR from respiratory secretions or blood within 48 h prior to assessment of eligibility.

ii. History of allergic reaction to blood or plasma products (as judged by the investigator).

iii. Medical conditions in which receipt of 500 mL intravascular volume may be detrimental to the patient (e.g., actively decompensated congestive heart failure).

iv. Enrollment in any other clinical trial for an investigational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2020-04-26 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-10-10 (Actual)

PRIMARY OUTCOMES:
Decrease length of stay | From date on which intervention given until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 1 month
  Decrease length of stay in hospital , Decrease length of stay in ICU/special care unit
Overall mortality | From date on which intervention given until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 1 month
  Status alive or death
Incidence of adverse events related to Convalescent Plasma transfusion | After receiving intervention (CP) till 24 hours
  Any adverse event after the transfusion of Convalescent plasma which include TRALI, TACO, allergic reaction, anaphylaxis.

SECONDARY OUTCOMES:
Ordinal scale | From date on which intervention given until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 1 month
  Modified from WHO scale. It includes clinical status of patient in terms of respiratory support needed.
Improvement in Laboratory Parameters: Serum Ferritin | From date on which intervention given until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 1 month
  Time to improvement in serum ferritin levels after intervention
Improvement in Laboratory Parameters: Procalcitonin | From date on which intervention given until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 1 month
  Time to improvement in serum Procalcitonin levels after intervention
Improvement in Laboratory Parameters: C-Reactive Protein | From date on which intervention given until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 1 month
  Time to improvement in C-Reactive protein levels after intervention
Improvement in Laboratory Parameters: D-Dimer | From date on which intervention given until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 1 month
  Time to improvement in D-Dimer levels after intervention
Improvement in Laboratory Parameters: Complete Blood count | From date on which intervention given until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 1 month
  Time to improvement in complete blood count after intervention
Chest X-Ray findings | From date on which intervention given until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 1 month
  Time to improvement in chest X-Ray findings after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Hasan, MBBS, FCPS, Principal Investigator — Aga Khan University Hospital, Karachi
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hung IF, To KK, Lee CK, Lee KL, Chan K, Yan WW, Liu R, Watt CL, Chan WM, Lai KY, Koo CK, Buckley T, Chow FL, Wong KK, Chan HS, Ching CK, Tang BS, Lau CC, Li IW, Liu SH, Chan KH, Lin CK, Yuen KY. Convalescent plasma treatment reduced mortality in patients with severe pandemic influenza A (H1N1) 2009 virus infection. Clin Infect Dis. 2011 Feb 15;52(4):447-56. doi: 10.1093/cid/ciq106. Epub 2011 Jan 19. PMID 21248066
- [Background] Arabi Y, Balkhy H, Hajeer AH, Bouchama A, Hayden FG, Al-Omari A, Al-Hameed FM, Taha Y, Shindo N, Whitehead J, Merson L, AlJohani S, Al-Khairy K, Carson G, Luke TC, Hensley L, Al-Dawood A, Al-Qahtani S, Modjarrad K, Sadat M, Rohde G, Leport C, Fowler R. Feasibility, safety, clinical, and laboratory effects of convalescent plasma therapy for patients with Middle East respiratory syndrome coronavirus infection: a study protocol. Springerplus. 2015 Nov 19;4:709. doi: 10.1186/s40064-015-1490-9. eCollection 2015. PMID 26618098
- [Background] Shen C, Wang Z, Zhao F, Yang Y, Li J, Yuan J, Wang F, Li D, Yang M, Xing L, Wei J, Xiao H, Yang Y, Qu J, Qing L, Chen L, Xu Z, Peng L, Li Y, Zheng H, Chen F, Huang K, Jiang Y, Liu D, Zhang Z, Liu Y, Liu L. Treatment of 5 Critically Ill Patients With COVID-19 With Convalescent Plasma. JAMA. 2020 Apr 28;323(16):1582-1589. doi: 10.1001/jama.2020.4783. PMID 32219428
- [Background] Robbins JB, Schneerson R, Szu SC. Perspective: hypothesis: serum IgG antibody is sufficient to confer protection against infectious diseases by inactivating the inoculum. J Infect Dis. 1995 Jun;171(6):1387-98. doi: 10.1093/infdis/171.6.1387. PMID 7769272